CLINICAL TRIAL: NCT00419783
Title: A Phase 1, Randomized, Multiple Dose, Double Blind, 5-way Crossover Study of the Electrocardiographic Effects of Bilastine in Healthy Adult Subjects
Brief Title: A Randomized, Multiple Dose, Double Blind, 5-way Crossover Study of the Electrocardiographic (ECG) Effects of Bilastine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 459-09; BILA-459/09; AA24101
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Allergic rhinitis; Urticaria
MeSH Terms: conditions — Rhinitis, Allergic; Urticaria | interventions — bilastine; Ketoconazole; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Bilastine 20 mg
  Interventions: Drug: bilastine
- 2 (Experimental): Bilastine 100 mg
  Interventions: Drug: Bilastine
- 3 (Active Comparator): Bilastine 20 mg + Ketoconazole 400 mg
  Interventions: Drug: Bilastine & Ketoconazole
- 4 (Active Comparator): Moxifloxacin 400 mg
  Interventions: Drug: Moxifloxacin
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bilastine — 20 mg tablets.
  Arms: 1
Drug: Bilastine — 100 mg (5 tablets of 20 mg)
  Arms: 2
Drug: Bilastine & Ketoconazole — 1 capsule containing bilastine 20 mg tablet + ketoconazole 400 mg tablet
  Arms: 3
Drug: Moxifloxacin — 1 capsule containing moxifloxacin 400 mg tablet
  Arms: 4
Drug: Placebo — Placebo tablets
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the effect of two doses of bilastine (20 and 100 mg) compared to bilastine 20 mg administered with ketoconazole 400 mg, moxifloxacin 400 mg, and placebo. Subjects will receive each of the five study treatments in a crossover fashion administered once daily for 4 days.

DETAILED DESCRIPTION:
This is a single center, Phase 1 study that utilizes a randomized, multiple-dose, double-blind, 5-way crossover design with a placebo control and two active controls. A minimum seven day washout period following four days of dosing for each of the five treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no clinically significant findings note on screening assessments including medical history, physical examination and laboratory results

Exclusion Criteria:

* Clinically significant medical condition
* Clinically significant history of ECG abnormalities or family history of QTc interval syndrome
* Use of tobacco and/or nicotine products >3 months prior to screening
* Use of any prescription medications within 14 days prior to screening
* Use of over the counter medications (including herbal products) within 7 days prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
QTc Interval prolongation | 4 days

SECONDARY OUTCOMES:
vital signs, adverse events, and routine clinical laboratory tests | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Allison, MD, Principal Investigator — MDS Pharma Services (US)
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States

REFERENCES:
- [Background] Church MK. Safety and efficacy of bilastine: a new H(1)-antihistamine for the treatment of allergic rhinoconjunctivitis and urticaria. Expert Opin Drug Saf. 2011 Sep;10(5):779-93. doi: 10.1517/14740338.2011.604029. Epub 2011 Aug 11. PMID 21831011
- [Result] Tyl B, Kabbaj M, Azzam S, Sologuren A, Valiente R, Reinbolt E, Roupe K, Blanco N, Wheeler W. Lack of significant effect of bilastine administered at therapeutic and supratherapeutic doses and concomitantly with ketoconazole on ventricular repolarization: results of a thorough QT study (TQTS) with QT-concentration analysis. J Clin Pharmacol. 2012 Jun;52(6):893-903. doi: 10.1177/0091270011407191. Epub 2011 Jun 3. PMID 21642470
- [Result] Graff C, Struijk JJ, Kanters JK, Andersen MP, Toft E, Tyl B. Effects of bilastine on T-wave morphology and the QTc interval: a randomized, double-blind, placebo-controlled, thorough QTc study. Clin Drug Investig. 2012 May 1;32(5):339-51. doi: 10.2165/11599270-000000000-00000. PMID 22393898